CLINICAL TRIAL: NCT00555698
Title: Feasibility, Safety and Efficacy of Deep Brain Stimulation of the Internal Capsule for Severe and Medically Refractory Major Depression
Brief Title: Feasibility, Safety and Efficacy of Deep Brain Stimulation for Depression
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Ali Rezai, MD (Other)
Collaborators: Medtronic (Industry); The Cleveland Clinic (Other)
Responsible Party: Sponsor-Investigator, Ali Rezai, MD, MD, Ohio State University
Organization: Ohio State University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 6577
Record Dates: First submitted 2007-11-07; First posted 2007-11-09 (Estimated); Last update posted 2017-03-28 (Actual); Status verified 2017-03

CONDITIONS: Depression
Keywords: DBS; Depression
MeSH Terms: conditions — Depression | interventions — Deep Brain Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- DBS (Experimental): DBS
  Interventions: Device: Deep Brain Stimulations for Depression

INTERVENTIONS:
Device: Deep Brain Stimulations for Depression — Deep Brain Stimulations for Depression

SUMMARY:
The purpose of this investigation is to obtain a preliminary indication of the feasibility, safety and efficacy of capsular deep brain stimulation (DBS) as a treatment for intractable depression. Also, to to learn about a new treatment for severe depression that has not improved enough despite long-term treatment with medications and behavior therapy. The new treatment is called deep brain stimulation, or DBS.

In DBS, thin wires are used to carry electric current to parts of the brain that are thought to be involved in producing depression symptoms. Two wires are implanted surgically, and attached to battery packs implanted under the skin of the new chest below your collar bone.

DETAILED DESCRIPTION:
This protocol proposes a pilot/feasibility clinical study of therapeutic benefits of ventral capsule/ventral striatum deep brain stimulation (DBS) as a treatment in ten patients with intractable major depression (MD). Conservative estimates place MD's prevalence at 2.6% to 5.5% in men and 6.0% to 11.8% in women. Most conservative studies estimate a 20% complete refractoriness to medical and psychotherapeutic regimens. Given the prevalence of major depression in the general population, over 3.5 million Americans would be expected to manifest refractory illness if all those with depression received treatment. Study subjects will have MD of disabling severity, intractable to prolonged treatment attempts with conventional medication and pschotherapies. They must also have had electroconvulsive therapy. These refractory patients would be candidates for a destructive/lesioning brain surgery such as a radiofrequency cingulotomy.

These MD patients are analogous to medically intractable Parkinson's disease and tremor patients who until recently underwent similar destructive surgeries such as a pallidotomy or thalamotomy. The use of DBS technology with its inherent advantage of being fully reversible and adjustable has become standard of care for these disabled patients. Studies have demonstrated improved safety and efficacy of DBS over lesioning.

Recently, DBS technology has been employed in the lesioning target of the anterior limb of the internal capsule for OCD. These preliminary studies in Europe and now the US, are demonstrating improved outcomes for refractory OCD patients with regard to their OC symptoms as well as depressed mood. This amelioration of mood provides the basis on which anterior internal capsule DBS may help major depression patients.

Based on this rationale, we believe that DBS is a viable therapeutic surgical option in this group of severely ill MD patients. The standard DBS stereotactic surgical techniques employed by the CCF team in hundreds of movement disorder patients will be used. The DBS electrodes will be implanted bilaterally in the anterior limb of the internal capsule and connected subcutaneously to subclavicular programmable pulse generators.

ELIGIBILITY:
Inclusion Criteria:

* Major depression, severe, unipolar type, diagnosed by Structured Clinical Interview for DSM-IV (SCID-IV), judged to be of disabling severity
* 24-item Hamilton Depression Rating Scale (HDRS) score of at least 21
* Global Assessment of Function (GAF) score of 45 or less.
* A recurrent (>4 episodes) or chronic (episode duration >2 years) course and a minimum of 5 years since the onset of the first depressive episode. Major impairment in functioning or potentially severe medical outcomes (repeated hospitalizations, serious suicidal or other self-injurious behavior).
* Failure to respond to:

  * adequate trials (>6 weeks at the maximum recommended or tolerated dose) of primary antidepressants from at least 3 different classes and;
  * adequate trials (>4 weeks at the usually recommended or maximum tolerated dose) of augmentation/combination of a primary antidepressant using at least 2 different augmenting/combination agents (lithium, T3, stimulants, neuroleptics, anticonvulsants, buspirone, or a second primary antidepressant) and;
  * an adequate trial of ECT (>6 bilateral treatments) and;
  * an adequate trial of individual psychotherapy (>20 sessions with an experienced psychotherapist).
* Age 18 - 55 years.
* Able to comply with the operational and administrative requirements of participation in the study.
* Able to give written informed consent.
* Either drug-free or on a stable drug regimen for at least 6 weeks at the time of entry into the study.
* Good general health.

Exclusion Criteria:

* Current or past nonaffective psychotic disorder.
* Any current clinically significant neurological disorder or medical illness affecting brain function, other than motor tics or Gilles de la Tourette syndrome.
* Any clinically significant abnormality on preoperative magnetic resonance imaging (MRI)
* Any surgical contraindications to undergoing DBS, including labeled contraindications for DBS and/or inability to undergo presurgical MRI (cardiac pacemaker, pregnancy, metal in body, severe claustrophobia), infection, coagulopathy, inability to undergo an awake operation, significant cardiac or other medical risk factors for surgery.
* Current or unstably remitted substance abuse.
* Pregnancy and women of childbearing age not using effective contraception.
* History of severe personality disorder.
* Imminent risk of suicide (based on the judgment of the investigators).
* Not able to comply with the operational and administrative requirements of participation in the study (based on the judgment of the investigators).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2004-01; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Montgomery-Asberg Depression Rating Scale (MADRS), Hamilton Depression Rating Scale (HDRS) | These scales are administered on each postoperative clinic visit. Visits occur monthly, except during the open continuation phase, when they occur every three months.

SECONDARY OUTCOMES:
Inventory for Depressive Symptoms, Self-report (IDS-SR), Clinical Global Impressions (CGI), Patient Global Impressions (PGI), Global Assessment of Functioning (GAF), Social and Occupational Function Assessment Scale (SOFAS), Quality of LIfe Enjoyment and | These measures will be obtained at baseline, at the end of the initial chronic phase (typically after three months of chronic stimultion), at the end of the open continuation phase (at two years into the study).

CONTACTS AND LOCATIONS:
Overall Officials: Ali Rezai, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic Foundation, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Greenberg BD, Malone DA, Friehs GM, Rezai AR, Kubu CS, Malloy PF, Salloway SP, Okun MS, Goodman WK, Rasmussen SA. Three-year outcomes in deep brain stimulation for highly resistant obsessive-compulsive disorder. Neuropsychopharmacology. 2006 Nov;31(11):2384-93. doi: 10.1038/sj.npp.1301165. Epub 2006 Jul 19. PMID 16855529